CLINICAL TRIAL: NCT00514852
Title: Safety and Efficacy of an Artificial Tear for the Treatment of Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AG9818-002
Record Dates: First submitted 2007-08-08; First posted 2007-08-10 (Estimated); Results first posted 2009-12-15 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-11

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Carboxymethylcellulose Sodium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Carboxymethylcellulose and Glycerin based artificial tear
  Interventions: Drug: Carboxymethylcellulose and Glycerin based artificial tear
- 2 (Active Comparator): Carboxymethylcellulose
  Interventions: Drug: Carboxymethylcellulose

INTERVENTIONS:
Drug: Carboxymethylcellulose and Glycerin based artificial tear — 1 to 2 drops into each eye as needed but at least twice daily
  Arms: 1
Drug: Carboxymethylcellulose — 1 to 2 drops into each eye as needed but at least twice daily
  Other Names: Refresh Plus
  Arms: 2

SUMMARY:
The efficacy, safety and acceptability of a new artificial tear in subjects with dry eye will be compared to a currently-available artificial tear

ELIGIBILITY:
Inclusion Criteria:

* Mild, moderate or Severe Symptoms of Dry Eye

Exclusion Criteria:

* Uncontrolled systemic disease
* Use of systemic medications affecting dry eye
* Pregnancy or planning a pregnancy
* Contact lens wear

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2007-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Carboxymethylcellulose Based Artificial Tear: 1 to 2 drops into each eye as needed but at least twice daily
Period: Overall Study
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Started | 157 | 159
Completed | 152 | 154
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear | Total
Number analyzed (Participants) | 157 | 159 | 316
Age, Customized [Number; unit: participants]
  <40 years | 18 | 15 | 33
  >=40 years | 139 | 144 | 283
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 125 | 245
  Male | 37 | 34 | 71

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Day 30 in Ocular Surface Disease Index© Questionnaire Score
Description: Ocular Surface Disease Index© Questionnaire Score is measured on 12 domains; a 5-point scale (0-4) for each domain. Sum of the domain scores is normalized to a severity scale of 0-100 (0 = no symptoms, 100 = maximum severity)
Time Frame: Change from baseline at Day 30
Population: Intent to Treat Population (Modified)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Number analyzed (Participants) | 147 | 154
Units on a scale
  Day 1 (Baseline) | 44 (18.1) | 45.2 (18.3)
  Day 7 | -12.6 (14.9) | -13.6 (17.8)
  Day 30 | -16.3 (16.4) | -16.6 (20.3)

2. Secondary Outcome: Change From Baseline at Day 30 in Schirmer Test, With Anesthesia
Description: Schirmer Test measures the rate of the secretion of tears
Time Frame: Change from baseline at Day 30
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: mm/5min
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Number analyzed (Participants) | 157 | 159
mm/5min
  Day 1 (Baseline) | 9.2 (7.2) | 8.6 (6.8)
  Day 7 | 1.2 (5.1) | 1.2 (5.6)
  Day 30 | 1.7 (6.9) | 1.8 (7.3)

3. Secondary Outcome: Change From Baseline at Day 30 in Tear Break-Up Time, With Fluorescein
Description: Measures the stability of tear film. The average of 3 measures.
Time Frame: Change from baseline at Day 30
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Number analyzed (Participants) | 157 | 159
seconds
  Day 1 (Baseline) | 4.3 (2.1) | 4.3 (2.0)
  Day 7 | 0.9 (2.3) | 0.9 (2.1)
  Day 30 | 1.1 (2.7) | 0.9 (2.4)

4. Secondary Outcome: Patient Acceptability Score (Dryness) at Day 30
Description: Dryness Severity Visual Analog Scale is measured on a 0-100 point scale (0 = could not be worse, 100 = none at all).
Time Frame: Day 30
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Number analyzed (Participants) | 157 | 159
Units on scale
  Day 1 (Baseline) | 47.4 (22.8) | 44.6 (20.5)
  Day 7 | 60.7 (21.1) | 57.7 (22.5)
  Day 30 | 63.3 (22.7) | 63.8 (22.8)

5. Secondary Outcome: Patient Acceptability Score (Vision) at Day 30
Description: Vision Quality Visual Analog Scale is measured on a 0-100 point scale (0 = very poor, has never been worse, 100 = excellent, has never been better).
Time Frame: Day 30
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Number analyzed (Participants) | 157 | 159
Units on a scale
  Day 1 (Baseline) | 56.8 (22.4) | 54.2 (21.6)
  Day 7 | 65.3 (17.8) | 62.6 (19.6)
  Day 30 | 65.4 (20.1) | 66.4 (19.4)

6. Post Hoc Outcome: Vision Subscale of the Ocular Surface Disease Index Questionnaire© at Day 30
Description: Vision subscale of the Ocular Surface Disease Index Questionnaire© is measured on 6 domains; a 5-point scale (0-4) for each domain. Sum of the domain scores is normalized to a severity scale of 0-100 (0 = no symptoms, 100 = maximum severity)
Time Frame: Day 30
Population: Intent to Treat Population (Modified)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Number analyzed (Participants) | 147 | 154
Units on a scale
  Day 1 (Baseline) | 37.6 (21.5) | 41.6 (21.6)
  Day 7 | 24.8 (20.0) | 26.9 (20.2)
  Day 30 | 22.8 (20.4) | 25.6 (22.4)

7. Post Hoc Outcome: Ocular Surface Staining With Fluorescein (Central Cornea) at Day 30
Description: Central staining score is based on modified Oxford Scheme measured on a scale of 0-5 (0= no staining, 5= most severe staining)
Time Frame: Day 30
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Number analyzed (Participants) | 157 | 159
Units on a scale
  Day 1 (Baseline) | 0.7 (0.8) | 0.8 (0.8)
  Day 7 | 0.5 (0.7) | 0.5 (0.7)
  Day 30 | 0.4 (0.6) | 0.4 (0.7)

8. Secondary Outcome: Change From Baseline at Day 30 in Ocular Surface (Corneal) Staining With Fluorescein
Description: Sum of corneal staining over 5 zones; each zone was measured on a modified Oxford Scheme of 0-5 (0=no staining, 5=most severe staining), with total score from 0-25 (0= no staining, 25 = most severe staining)
Time Frame: Change from baseline at Day 30
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Number analyzed (Participants) | 157 | 159
Units on a scale
  Day 1 (Baseline) | 4.0 (3.3) | 4.4 (3.4)
  Day 7 | -1.2 (2.3) | -0.9 (2.4)
  Day 30 | -1.3 (2.4) | -1.5 (2.5)

9. Secondary Outcome: Change From Baseline at Day 30 in Ocular Surface (Conjunctival) Staining With Fluorescein
Description: Sum of conjunctival staining over 6 zones; each zone was measured on a modified Oxford Scheme of 0-5 (0=no staining, 5=most severe staining), with total score from 0-30 (0=no staining, 30=most severe staining)
Time Frame: Change from baseline at Day 30
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Number analyzed (Participants) | 157 | 159
Units on a scale
  Day 1 (Baseline) | 4.9 (4.4) | 5.1 (5.0)
  Day 7 | -1.1 (3.1) | -1.0 (3.2)
  Day 30 | -1.7 (3.3) | -1.5 (2.8)

10. Secondary Outcome: Change From Baseline at Day 30 in Subjective Evaluation of Symptom of Dryness Score
Description: Measures dry eye severity on a scale of 0-4 (0 = none, 4 = severe)
Time Frame: Change from baseline at Day 30
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Number analyzed (Participants) | 157 | 159
Units on a scale
  Day 1 (Baseline) | 2.8 (0.7) | 2.8 (0.8)
  Day 7 | -0.5 (0.8) | -0.5 (0.8)
  Day 30 | -0.7 (1.0) | -0.7 (0.9)

ADVERSE EVENTS:
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Serious Adverse Events (participants affected / at risk) | 1/157 | 1/159
Other Adverse Events (participants affected / at risk) | 0/157 | 0/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboxymethylcellulose and Glycerin Based Artificial Tear (N=157) | Carboxymethylcellulose Based Artificial Tear (N=159)
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.